CLINICAL TRIAL: NCT01463605
Title: Nimotuzumab Combined With Radiotherapy for Older Patients With Esophageal Cancer: a Single, Non-control Phase II Clinical Trial
Brief Title: Nimotuzumab Combined With Radiotherapy for Older Patients With Esophageal Cancer: a Single, Non-control Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Liang Jun, Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-49/484
Record Dates: First submitted 2011-10-30; First posted 2011-11-02 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Esophageal Cancer
Keywords: radiotherapy; targeted therapy; esophageal cancer; older
MeSH Terms: conditions — Esophageal Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiotherapy (Other): It is just a single group assignment
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 200mg,once per week,for 5 to 6 weeks

SUMMARY:
For patients who are unable to receive surgery or having local advanced esophageal cancer stages, concurrent chemoradiotherapy is recommended. But radiotherapy is the main strategy for older patients because of their chemoradiotherapy intolerance. The whole world focused on targeted therapy which has strong specialties and mild toxicities. So combined targeted therapy and radiotherapy may be a novel strategy for older patients with esophageal cancer. Nimotuzumab is a EGFR monoclonal antibody. This clinical trial is to study the effect and safety of Nimotuzumab in combined with radiotherapy for older patients with esophageal cancer. All patients receive intensity modulated radiotherapy with conventional fraction. Nimotuzumab with 200mg is given weekly for all patients during radiotherapy.

DETAILED DESCRIPTION:
Study Design Primary Purpose: To evaluate the response rate, progression-free survival, overall survival and complications.

Study Phase: Phase II Intervention Model: Targeted therapy combined with radiotherapy Number of Arms: One Masking: No Allocation: 30 patients for one single group Enrollment: 30 patients

Eligibility Criteria Inclusion Criteria: 1. ≥ 70 year-old, 2. Thoracic segment esophageal cancer with stage II to IV (supraclavicular lymph node metastasis only), 3. No previous surgery, radiotherapy or chemotherapy of cancer was allowed, 4. Estimated survival time ≥ 3 months, 5. KPS > 60, 6. No serious diseases of important organs, 7. Signed consent forms voluntarily.

Exclusion Criteria: 1. Psychopath, 2. History of other malignant disease which has not been cured, 3. Joining other clinical trial prior this study.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 70 years or older;
2. treatment naive patients with histologically proven thoracic-segment EC that was inoperable and who could not tolerate CCRT;
3. stage II-IV disease (supraclavicular lymph node metastasis only), according to the 6th American Joint Committee on Cancer TNM staging system;
4. estimated survival time ≥3 months;
5. Karnofsky performance score ≥70;
6. adequate bone marrow, as well as hepatic and renal function;
7. voluntary written consent provided prior to treatment.

Exclusion Criteria:

1. esophagobronchial or esophagomediastinal fistula;
2. patients who had joined other clinical trials prior to this treatment;
3. serious heart, liver, and/or kidney insufficiency;
4. serious infectious disease;
5. relapse disease or distant metastasis;
6. recently diagnosed neoplastic diseases;
7. previous receipt of surgery, chemotherapy, or radiotherapy for EC.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Safety of Nimotuzumab combined with Radiotherapy for older patients | 2 years
  To observe the adverse events during the treatment

SECONDARY OUTCOMES:
Efficacy of Nimotuzumab combined with Radiotherapy for older esophageal cancer patients | 3 years
  To observe the response rate, progress-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Liang Jun, Doctor, Principal Investigator — Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- See also: This review discuss pre-clinical data and the rationale for targeting these pathways and summarize the results of clinical trials to-date. — http://www.elsevierhealth.com/journals/ctrv
- See also: Changing healthcare practice of older adults with late-stage non-small cell lung cancer: practical considerations of targeted therapy in primary care and oncology. — http://www.ncbi.nlm.nih.gov/sites/entrez